CLINICAL TRIAL: NCT06561893
Title: Effect of L. Plantarum Probiotic Supplementation on Broccoli Sulforaphane Bioavailability: Randomised Double-blind Placebo-controlled Crossover Study
Acronym: PRO-BROC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: The University of Queensland (Other); PepsiCo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 6190780
Record Dates: First submitted 2024-06-18; First posted 2024-08-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Nutrition, Healthy
Keywords: broccoli; sulforaphane; probiotic; gut microbiota; L. plantarum; bioavailability; cross-over trial

STUDY DESIGN:
Intervention Model Description: Randomised Double-blind Placebo-controlled Crossover Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (L. plantarum) supplementation (Active Comparator): Dose: 20 Billion CFU/day for 14 days (total of two pills of 10 Billion CFU)
  Interventions: Dietary Supplement: Broccoli sprouts extract supplementation
- Placebo (dextrose) supplementation (Placebo Comparator): Dose: 700 mg of dextrose (total of two pills; 2 x 350 mg pills)
  Interventions: Dietary Supplement: Broccoli sprouts extract supplementation

INTERVENTIONS:
Dietary Supplement: Broccoli sprouts extract supplementation — Intake of broccoli sprouts extract supplement (Brand: Source Naturals, Scotts Valley, CA 95066 - USA) in an acute dose (84 umol of glucoraphanin) before and after 2 weeks of probiotic or placebo supplementation, to assess sulforaphane bioavailability measured in urine metabolites

SUMMARY:
Broccoli has the precursor of an active compound (sulforaphane) that has shown a wide range of health promoting benefits. Sulforaphane formation depends on the conversion of glucoraphanin (precursor) by myrosinase enzyme. Thus, the bioavailability of sulforaphane is affected by myrosinase activity. Some bacteria, such as L. plantarum (probiotic), have shown they can also convert glucoraphanin to sulforaphane in vitro. This study investigates the effect of short-term L. plantarum supplementation on broccoli sulforaphane bioavailability in humans using a randomised double-blind placebo-controlled crossover trial.

DETAILED DESCRIPTION:
Brassicas (i.e. broccoli, kale, cabbage) are a group of edible plants that contain a phytochemical called glucoraphanin that upon enzymatic hydrolysis forms the bioactive form sulforaphane. Sulforaphane has shown consistent in vitro and in vivo (animals) anti-cancer activity. The enzyme responsible for this conversion is called myrosinase; however, the enzymatic activity of myrosinase can be affected by several biological factors (e.g. plant variety, growth conditions, etc...) and food processing (e.g. cooking, drying, etc...). Broccoli is one of the richest sources of glucoraphanin, but its myrosinase activity can be easily lost during cooking: 10 minutes at 70 °C reduces the enzyme activity by 95%. This means broccoli prepared this way will contain little to no biologically active sulforaphane. Therefore, is important to find strategies to increase the bioavailability of sulforaphane in broccoli and other brassicas for human consumption.

Certain bacteria have shown myrosinase-like activity and were able to convert glucoraphanin to sulforaphane in vitro, one of these bacteria is Lactiplantibacillus plantarum. This bacterium is present in the human gut, however, there is a large biological variability in the prevalence of this bacteria between individuals. Several human studies have demonstrated that chronic (>1 week) consumption of probiotic supplements containing L. plantarum was able to increase the presence of this bacterium in human gut participants. Thus, the investigators aim to test if supplementing participants with L. plantarum will increase the bioavailability of sulforaphane, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults (male and female)
* age range of 18-65 years
* BMI range of 18-30 kg/m2

Exclusion Criteria:

* have been on a course of antibiotics within the period of the past 3 months.
* have allergies or intolerance towards probiotic substances or broccoli used in the study and/or food intolerances associated with gastrointestinal upset.
* have been taking pre- or probiotics supplements regularly during the last month prior (this does not include foods containing probiotics and/or prebiotics foods)
* are following any restricting diet (e.g., vegan, FODMAP, etc.).
* have a gastrointestinal inflammatory condition (e.g., irritable bowel syndrome, inflammatory bowel diseases, coeliac diseases, constipation, etc.).
* have a medical condition or take medication for any heart, endocrine, or metabolic condition, such as high blood pressure, high cholesterol, insulin resistance, or diabetes, or autoimmune disease.
* are a pregnant and/or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Bioavailability of sulforaphane | From baseline to the end of each condition at 2 weeks, followed by 2 weeks of wash-out, and before and after the next condition
  Bioavailability (%) of sulforaphane (will be estimated by dividing the cumulative amount of sulforaphane mercapturic acid excreted in urine in 24 h by the consumed amount of glucoraphanin (Vermeulen et al., 2008)) before and after chronic consumption of L. plantarum compared with placebo.

SECONDARY OUTCOMES:
Sulforaphane pharmacokinetics: Area under the curve | From baseline to the end of each condition at 2 weeks, followed by 2 weeks of wash-out, and before and after the next condition.
  Measurement of the definite integral of the concentration of sulforaphane (and its metabolites) in blood plasma as a function of time.
Sulforaphane pharmacokinetics: Cmax | From baseline to the end of each condition at 2 weeks, followed by 2 weeks of wash-out, and before and after the next condition.
  Measurement of the maximum plasma concentration (Cmax) of sulforaphane (and its metabolites) indicating the value of the highest concentrations reached in the plasma.
Sulforaphane pharmacokinetics: Tmax | From baseline to the end of each condition at 2 weeks, followed by 2 weeks of wash-out, and before and after the next condition.
  Measurement of the time taken for sulforaphane (and its metabolites) to reach the maximum concentration (Cmax) after administration of the supplement that needs to be absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Torquati, PhD, Principal Investigator — University of Exeter
Locations (2):
- United Kingdom (2):
  - The Department of Public Health and Sport Sciences, University of Exeter Medical School, Faculty of Health and Life Sciences, University of Exeter, Exeter, Devon
  - Richard's Building, St Luke's Campus, Exeter, Devon

IPD SHARING:
Plan to Share IPD: No
Participant details (name, age, sex, etc.) will be stored in a password secured as per university guidelines. Participants will be allocated a code (ID number) at enrolment, and this will be used to refer to them hereafter. Data will be collected and entered under a participant's ID number, and analysed and stored as such. Only researchers listed in this application will have access to all data. Presentations, reports and publications will only include aggregated data with no personal or individual data included. Anonymised databases will be made available upon request or deposit in open repository upon request of journal.

REFERENCES:
- [Background] Oloyede OO, Wagstaff C, Methven L. The Impact of Domestic Cooking Methods on Myrosinase Stability, Glucosinolates and Their Hydrolysis Products in Different Cabbage (Brassica oleracea) Accessions. Foods. 2021 Nov 24;10(12):2908. doi: 10.3390/foods10122908. PMID 34945460
- [Background] Gonzalez F, Quintero J, Del Rio R, Mahn A. Optimization of an Extraction Process to Obtain a Food-Grade Sulforaphane-Rich Extract from Broccoli (Brassica oleracea var. italica). Molecules. 2021 Jul 1;26(13):4042. doi: 10.3390/molecules26134042. PMID 34279379
- [Background] Iahtisham-Ul-Haq, Khan S, Awan KA, Iqbal MJ. Sulforaphane as a potential remedy against cancer: Comprehensive mechanistic review. J Food Biochem. 2022 Mar;46(3):e13886. doi: 10.1111/jfbc.13886. Epub 2021 Aug 5. PMID 34350614
- [Background] Surono IS, Simatupang A, Kusumo PD, Waspodo P, Verbruggen S, Verhoeven J, Venema K. Effect of Different Functional Food Supplements on the Gut Microbiota of Prediabetic Indonesian Individuals during Weight Loss. Nutrients. 2022 Feb 13;14(4):781. doi: 10.3390/nu14040781. PMID 35215431
- [Background] Ye JH, Huang LY, Terefe NS, Augustin MA. Fermentation-based biotransformation of glucosinolates, phenolics and sugars in retorted broccoli puree by lactic acid bacteria. Food Chem. 2019 Jul 15;286:616-623. doi: 10.1016/j.foodchem.2019.02.030. Epub 2019 Feb 14. PMID 30827654
- [Background] Cai YX , Augustin MA , Jegasothy H , Wang JH , Terefe NS . Mild heat combined with lactic acid fermentation: a novel approach for enhancing sulforaphane yield in broccoli puree. Food Funct. 2020 Jan 29;11(1):779-786. doi: 10.1039/c9fo02089f. PMID 31922158
- [Background] Vermeulen M, Klopping-Ketelaars IW, van den Berg R, Vaes WH. Bioavailability and kinetics of sulforaphane in humans after consumption of cooked versus raw broccoli. J Agric Food Chem. 2008 Nov 26;56(22):10505-9. doi: 10.1021/jf801989e. PMID 18950181